CLINICAL TRIAL: NCT00364702
Title: Virtual Reality a Novel Screening and Treatment Aid in Attention Deficit Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 45/04
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2006-07

CONDITIONS: ADHD
Keywords: Virtual Reality; ADHD; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate

SUMMARY:
Using a virtual reality program in screening and treatment of ADHD.

DETAILED DESCRIPTION:
Virtual Reality is a novel program designed to imitate a real classroom environment including various distractions. It includes a head monitor to track eye movements Children aged 10-20 years with ADHD will use the program with and without methylphenidate(1 mg/kg). Their results will be compared to a control group.

Parental consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ADHD-DSM4 criteria AGE 10-20 YEARS normal neurological examination IQ>80

Exclusion Criteria:

ABNORMAL NEUROLOGICAL STATUS

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Virtual Reality program test results

CONTACTS AND LOCATIONS:
Overall Officials: V. Gross, Prof/ md, Study Chair — Shaari Zedek Pediatric Neurology Unit
Locations (1):
- Shaari Zedek Pediatric Neurology Unit, Jerusalem, Israel